CLINICAL TRIAL: NCT07072754
Title: Effectiveness of Yoga and Combined Exercise in Female With Rheumatoid Arthritis: Randomized Controlled Trial
Brief Title: Effectiveness of Yoga and Combined Exercise in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Sevtap Günay, Associate Professor Doctor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rheumatoid Arthritis and Yoga
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: rheumatoid arthritis; yoga; combined exercise; pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Mind-Body Therapies; Yoga; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga (Experimental): The yoga program, led by a physiotherapist who is also a certified yoga instructor , with two sessions per week lasting one hour each. It was applied for a total of 8 weeks.
  Interventions: Other: Mind-body therapy
- Combined Exercise (Experimental): Patients in the exercise group were given a program that included warm-up, low-impact aerobic, strengthening, and cooling phases, totaling 60 minutes, repeated twice a week for eight weeks.
  Interventions: Other: Exercise
- Control (No Intervention): No exercise was applied to the subjects included in the control group.

INTERVENTIONS:
Other: Mind-body therapy — The yoga program, led by a physiotherapist who is also a certified yoga instructor , with two sessions per week lasting one hour each. Foam yoga blocks, belts, and armless chairs were also available in the classes, where the participants were to support compliance with the program. The yoga program was planned as 10 minutes of centering and breathing practice, 10 minutes of warm-up practice, 30 minutes of supine, standing, sitting, prone, and supine yoga postures, and 10 minutes of relaxation. New postures were introduced every two weeks as the program progressed. After the eight-week session, the participants were encouraged to continue the program at home twice a week
  Other Names: Yoga
  Arms: Yoga
Other: Exercise — Patients in the exercise group were given a program that included warm-up, low-impact aerobic, strengthening, and cooling phases, totaling 60 minutes, repeated twice a week for eight weeks. Aerobic exercise was performed by standing still for 25 minutes at moderate intensity based on perceived effort. Strengthening exercises included one set of 10 repetitions for each movement. Exercises were progressed according to the modified Borg's scale. Strengthening exercises included core muscles such as the deltoid, abdominals, quadriceps femoris, and hamstrings and were performed using body weight or elastic resistance bands
  Arms: Combined Exercise

SUMMARY:
This study aims to elucidate the potential benefits of exercise for individuals with rheumatoid arthritis. The findings are expected to contribute to the development of novel and effective therapeutic approaches, ultimately leading to an improved quality of life for patients. For both patients and healthcare professionals, a clearer understanding of exercise's role in rheumatoid arthritis management will serve as a crucial guide in formulating individualized treatment plans. The results of our study will provide valuable insights to aid in developing strategies aimed at enhancing the physical and mental well-being of individuals afflicted with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that significantly impacts daily life by causing pain, swelling, and restricted movement in the joints. This study aimed to investigate the effects of yoga and combined exercise methods on the symptoms of RA in individuals with the condition, comparing them to a control group that did not engage in exercise. Participants were comprehensively evaluated at baseline, week 8, and week 20 for key variables such as pain level, balance, joint mobility, depression level, fatigue level, and quality of life. This research seeks to reveal the potential benefits of exercise in RA management, thereby contributing to the development of effective treatment approaches that improve patients' quality of life. The findings will help both patients and healthcare professionals better understand the role of exercise in RA treatment, serving as a crucial guide for creating individualized treatment plans. The results are expected to offer valuable insights for developing strategies to enhance the physical and mental health of individuals with RA.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of RA for at least six months according to the ACR criteria
* aged between 18-65 years,
* under stabil medications at least four weeks
* the disease activity score 28 (DAS 28) <2.6 (Remission period) of each patient at least three months
* ability to provide written informed consent.

Exclusion Criteria:

* had pain that prevents general mobility,
* had neurologic, cardiologic (arrhythmias, myocardial infarction, uncontrolled metabolic disease,
* known electrolyte abnormalities,
* systolic BP > 200 mm Hg or diastolic BP > 115 mm Hg)
* respiratory pathology,
* pregnancy
* had malignancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 74 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | From enrollment to the end of treatment at 8 weeks and 20 weeks after baseline
  The Visual Analogue Scale (VAS) was used for pain intensity assessment in all patients. The scale is a 10-cm line, with the leftmost part showing no pain and the rightmost part showing maximum pain. Patients were asked to point to the proper place on the line according to the pain they experienced last week. An increase of 20% or above indicates clinical significance in VAS.

SECONDARY OUTCOMES:
Balance Index | From enrollment to the end of treatment at 8 weeks and 20 weeks after baseline
  The Berg Balance Scale (BBS) was used to evaluate the functional balance status. It is a 14-item test of functional balance. Each item is scored between 0-4, with a maximum score of 56. Higher scores represent a good balance level. It assesses static balance during standing and sitting and dynamic balance during walking. The Turkish validity and reliability of the scale were conducted by Sahin et. al.
Mobility Level | From enrollment to the end of treatment at 8 weeks and 20 weeks after baseline
  The Timed Up and Go test (TUG) was also used to evaluate the balance and mobility of the patients. This test is used to measure walking speed and evaluate balance, physical mobility, and the ability to go outside alone. For the TUG test, patients were asked to stand up from a chair with armrests, to walk 3 meters, to turn and walk back to the chair, and to sit down again to the chair. The time it took to complete the test was recorded using the electronic stopwatch. The minimum clinical significance of TUG was given as a decrease of 1.14 seconds.
Depression Level | From enrollment to the end of treatment at 8 weeks and 20 weeks later baseline
  The severity of depression was evaluated using the Beck Depression Inventory Scale (BDI), which has 21 items and a total score of 63. The cut-off scores for the RA population revealed 0-12 for minimal, 13-18 for mild, 19-28 for moderate, and 29-63 for severe depression. The Turkish validity and reliability of the scale were conducted by Hisli et. al..
Fatigue Level | From enrollment to the end of treatment at 8 weeks and 20 weeks later baseline
  The Fatigue Severity Scale (FSS) was used to measure the impact of fatigue on patients. It contains nine statements, rated on a Likert scale of 1 to 7, where 1 indicates completely disagree, and 7 indicates agree entirely. Higher scores indicate higher fatigue levels. In a study conducted on systemic lupus patients, the minimum clinical significance of FSS was given as a decrease of 0.6 points or more. The Turkish validity and reliability of the scale were conducted by Gencay-Can.
Quality of Life Level | From enrollment to the end of treatment at 8 weeks and 20 weeks later baseline
  Short Form 36 (SF-36) was used to assess health-related quality of life. The SF-36 is a widely applied generic instrument for measuring health status and consists of eight dimensions: physical functioning, social functioning, physical role, emotional role, mental health, vitality, bodily pain, and general health perceptions. Scores range from 0 (worst) to 100 (best), with higher scores indicating better health status. The Turkish validity and reliability of the scale were conducted by Bilir Kaya et. al.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Umay Altas, Associate Professor Doctor, Principal Investigator — Izmir Bakircay University
Locations (1):
- Katip Celebi University Atatürk Education and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal data will not be shared. All data will be shared blindly by special request, provided that a valid reason is given.